CLINICAL TRIAL: NCT06326099
Title: A Mobile-Based Intervention to Address Heavy Drinking and Binge Eating in College Students
Brief Title: Brief Binge Eating and Drinking Online Intervention
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern California (Other)
Responsible Party: Principal Investigator, Eric Pedersen, Associate Professor, University of Southern California
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R34AA030655 (NIH)
Record Dates: First submitted 2024-03-15; First posted 2024-03-22 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-03

CONDITIONS: Binge Eating; Binge Drinking
MeSH Terms: conditions — Bulimia; Binge Drinking

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Brief Online Binge Eating and Drinking Intervention (Experimental): The intervention is a 30 minute mobile phone program designed to address binge eating and drinking. The program addresses underlying loss of control, impulsivity, and emotion regulation common to both binge drinking and binge eating through videos, interactive activities, and psychoeducation.
  Interventions: Behavioral: Brief Online Binge Eating and Drinking Intervention
- Resources Only (No Intervention): Campus-specific resources for how to access the university's counseling office (i.e., student mental health services), information about the Eating Disorders program at the university, and information on accessing the university's alcohol and drug awareness offices.

INTERVENTIONS:
Behavioral: Brief Online Binge Eating and Drinking Intervention — The intervention is an online mobile phone program developed by our research team. It builds upon efficacious brief alcohol interventions with college students by addressing underlying loss of control, impulsivity, and emotion regulation through the use of videos, interactive activities, and psychoeducation.
  Other Names: Sip n' Savor
  Arms: Brief Online Binge Eating and Drinking Intervention

SUMMARY:
This pilot project targets both binge drinking and binge eating behavior in college students through a mobile-based online program that provides students with evidence-based intervention material designed to reduce the incidence of both behaviors and encourage students to seek more formal in-person counseling.

DETAILED DESCRIPTION:
Despite the prevalence of binge drinking and binge eating behaviors among college students, few students seek care for either. Intervening with college students early is essential as untreated symptoms of binge drinking and binge eating behaviors can become more severe and persistent over time, often leading to diagnosed disorders and lasting consequences on students' social functioning, physical health, and educational attainment. Thus, the major goal of this research study is to target both binge drinking and binge eating behavior in college students through a mobile-based online program that provides students with evidence-based intervention material designed to reduce the incidence of both behaviors, as well as encourage students to seek more formal in-person counseling. The intervention combines two innovations to facilitate behavior change: (1) personalized drinking and binge eating intervention content with harm reduction and cognitive behavioral skills proven to be efficacious in reducing these problematic behaviors among college students delivered via (2) a mobile-based program that increases accessibility, is easy and engaging to use, and broadens the accessibility of the intervention content to an often non-treatment seeking group. The intervention is informed by evidence-based practices, with student and expert feedback, to help limit alcohol consumption, engage in healthier eating behaviors, and practice alternate strategies to manage negative affect.

ELIGIBILITY:
Inclusion Criteria:

* full time undergraduate student at the study site
* between the ages of 18 and 24
* ability to speak and read English
* at least two occasions of binge drinking (5 or more drinks in a row for males, 4 (i.e., an objectively large amount of food with a self-reported loss of control) in the past 28 days
* at least two occasions of binge eating (i.e., an objectively large amount of food with a self-reported loss of control)151 in the past 28 days
* no receipt of mental health or substance use care in the past month.

Exclusion Criteria:

* not meeting eligibility criteria

Ages: 18 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 300 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Frequency of past 28-day binge drinking | Baseline, one-month follow-up, and three-month follow-up
  Number of binge drinking episodes in the past 28 days
Frequency of past 28-day binge eating | Baseline, one-month follow-up, and three-month follow-up
  Number of binge eating episodes in the past 28 days
Brief Young Adult Alcohol Consequences Questionnaire (B-YAACQ) | Baseline, one-month follow-up, and three-month follow-up
  21 alcohol-related consequences experienced in the past month. Sum positive responses to get a score from 0 to 24 (higher score indicates greater number of consequences)

SECONDARY OUTCOMES:
Mental Health/Substance Use Disorder Treatment History Inventory | Baseline, one-month follow-up, and three-month follow-up
  Utilization of mental health and/or substance use care

IPD SHARING:
Plan to Share IPD: Yes
Following the NIH Data Sharing Policy and Implementation Guidelines, we plan to make the datasets available for sharing at the time that the main project findings are accepted for publication during the final year of the project.
Supporting Information: Study Protocol
Time Frame: Within one year of the main effects paper being submitted for publication
Access Criteria: Individual researchers can contact the PIs for data and through filling out a data request and use form that we will create for the purposes of data sharing.